CLINICAL TRIAL: NCT02320409
Title: A Food Effect Phase I Study of the Sulfatinib in Healthy Subjects
Brief Title: A Food Effect Phase I Study of the Sulfatinib in Healthy Subjects (HMPL-012)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-012-00CH2
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Healthy
Keywords: Subjects
MeSH Terms: interventions — surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sulfatinib ,after general diet (Experimental): First cycle, single oral Sulfatinib after general diet intake; Second cycle, Sulfatinib before general diet intake.
  Interventions: Drug: Sulfatinib
- Sulfatinib, before general diet (Experimental): First cycle, single oral Sulfatinib before general diet intake;Second cycle,single oral Sulfatinib after general diet intake
  Interventions: Drug: Sulfatinib

INTERVENTIONS:
Drug: Sulfatinib — 250mg Sulfatinib ,single dose,oral
  Other Names: HMPL-012

SUMMARY:
The purpose of this study is to evaluate to determine the effect of food on the PK of a single dose of 250 mg Sulfatinib and its metabolites in healthy subjects.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate to determine the effect of food on the PK( pharmacokinetics) of a single dose of 250 mg Sulfatinib and its metabolites in healthy subjects and to assess the safety and tolerability of single doses of 250mg in healthy subjects.This study will be an open-label, randomized, two-period, crossover PK food effect study of Sulfatinib administered orally at 250 mg. Subjects will be screened for eligibility up to 14 days prior to entry into the study,there will be 2 treatments,2 weeks follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Males , between 18 and 55 years of age, inclusive.
* Body mass index (BMI) within the range of 20 to 30 kg/m2, inclusive.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, and vital signs.
* Adequate hepatic, renal, heart, and hematologic functions
* Male subjects who are either sterile or agree to use and get the agreement of their sexual partners to use , during the period from informed consent until 90 days following Study Completion, 1 of the following approved methods of contraception: condom, use by female sexual partner of an intrauterine device, contraceptive sponge, diaphragm, or use of a cervical cap; or an oral, implantable, transdermal, injectable contraceptives or other contraceptive measures.
* Able to comprehend and willing to sign an informed consent form (ICF).

Exclusion Criteria:

* disease history or clinical manifestation of any significant metabolic/endocrine, allergic, dermatological, hepatic, renal, hematological, pulmonary, immune, cardiovascular, gastrointestinal, genitourinary, neurological, or psychiatric disorder(as determined by the Investigator).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator.
* serum total bilirubin>34.2 umol/L；
* serum albumin<35 g/L；
* GFR < 80 mL/min/1.73m2. Algorithm: GFR (mL/min/1.73m2) =186 × (SCr)-1.154 × (Age)-0.203, Scr= serum creatinine, mg/dL；
* Blood pressure greater than 140/90.
* History or presence of an abnormal ECG, which, in the Investigator's opinion, is clinically significant.
* Smoking more than 10 cigarettes daily without intention to quit smoking during study.
* History of stomach or intestinal surgery, nephrectomy, cholecystectomy or resection that would potentially alter absorption and/or excretion of orally administered drugs as determined by the investigator (appendectomy and/or hernia repair may be allowed).
* Significant allergy history(eg. drug allergy); acute allergic rhinitis or food allergy within 2 weeks prior to informed consent.
* Donation of blood or plasma ≥ 500 mL from 30 days prior to informed consent, or of blood or plasma ≥250 mL from 2 weeks prior to informed consent.
* Receipt of blood products within 2 months prior to informed consent;
* Poor peripheral venous access.
* Participants who are positive for hepatitis B surface antigen (HBs antigen) or hepatitis B core antibody , hepatitis C virus (HCV) antibody;
* Participants who are human immunodeficiency virus (HIV)-positive;
* Diagnosis of alcoholism or drug addiction within 1 year prior to informed consent.
* Participation in any other investigational drug study in which receipt of an investigational study drug occurred within 5 half-lives or 28 days, whichever is longer prior to informed consent.
* Use of any prescription medications or products within 14 days prior to informed consent.
* Use of any over-the-counter (OTC), non-prescription preparations (including vitamins, minerals, and phytotherapeutic, herbal,) within 7 days prior to informed consent.
* Use of alcohol-, grapefruit-, Seville orange-, or caffeine-containing foods, juices, or beverages within 72 hours prior to informed consent.
* Use of known hepatic or renal clearance altering agents (eg, erythromycin, cimetidine, barbiturates, phenothiazines, or herbal/plant derived preparations such as St. John's Wort, etc.) for a period of 60 days prior to first dose;
* principal investigator, investigator, pharmacist, Clinical Research Coordinator or any personnel related to this study.
* Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-12; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The following PK parameters will be derived from the plasma concentration-time profile of Sufatinib following administration | 1-3 days
  Area Under Curve (AUC), both from time zero to time with last observation and from time zero to infinity;;Maximum plasma concentration (Cmax);Time to reach the Cmax (Tmax);elimination half-life

SECONDARY OUTCOMES:
AE (adverse event) will be summarized by type and severity | 1 day to the 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Chen Yu, Dr., Principal Investigator — Xuhui Center Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Qian H, Wu X, Chen Q, Li T, Wang W, Jia J, Yu C, Li K, Sai Y, Su W, Liu Y. Effects of Food on the Pharmacokinetic Properties of Surufatinib: A Phase I, Single-dose, Randomized, Open-label Crossover Study in Healthy Subjects. Clin Ther. 2020 Sep;42(9):1778-1786. doi: 10.1016/j.clinthera.2020.07.010. Epub 2020 Aug 13. PMID 32800383